CLINICAL TRIAL: NCT04935762
Title: A Phase II, Randomized, Placebo-Controlled, Double-Blind, Crossover Study to Evaluate the Use of CST-103 Co-administered With CST-107 on Freezing of Gait in Subjects With Parkinson's Disease
Brief Title: A Study of CST-103 Co-administered With CST-107 in Subjects With Parkinson's Disease Having Freezing of Gait (CLIN-012)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: CuraSen Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CST103/CST107-CLIN-012
Record Dates: First submitted 2021-06-09; First posted 2021-06-23 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Freezing of Gait Symptoms in Parkinson's Disease

STUDY DESIGN:
Intervention Model Description: Two 14-day periods, 2-way crossover design
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-Blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CST-103/CST-107 to Placebo (Experimental): Subjects will receive daily doses of CST-103 co-administered with CST-107 for 14 days, followed by a washout period of no drug for 14 days, followed by matching placebo for CST-103 and matching placebo for CST-107 for 14 days.
  Interventions: Drug: CST-103, CST-107, matching placebo
- Placebo to CST-103/CST-107 (Experimental): Subjects will receive daily doses of matching placebo for CST-103 and matching placebo for CST-107 for 14 days, followed by a washout period of no drug for 14 days, followed by daily doses of CST-103 co-administered with CST-107 for 14 days.
  Interventions: Drug: CST-103, CST-107, matching placebo

INTERVENTIONS:
Drug: CST-103, CST-107, matching placebo — CST-103 and matching placebo orange capsules; CST-107 and matching placebo white capsules

SUMMARY:
This is a Phase II, randomized, placebo-controlled, double-blind, crossover study to evaluate the effect of multiple oral doses of CST-103 in the presence of CST-107 on Freezing of Gait (FOG) symptoms in subjects with Parkinson's Disease (PD).

DETAILED DESCRIPTION:
Approximately 25 PD subjects with FOG symptoms will be enrolled in a 2 period, 2-way crossover design following study eligibility confirmation during the screening period.

During each treatment period, subjects will receive daily doses of CST-103 co-administered with CST-107 or matching placebo for 14 days. Each treatment period will be separated by a washout period of at least 14 days.

All subjects will complete clinical and pharmacodynamic assessments during each treatment period. Pharmacokinetic blood samples will be collected prior to and after study medication administration. Pharmacodynamic blood samples will also be collected to investigate the effects of CST-103 co-administered with CST-107 on inflammatory and neurodegenerative biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects ≥ 30 and ≤ 80 years of age, at time of informed consent.
* Diagnosed with Parkinson's Disease, as defined by the United Kingdom Parkinson Disease Brain Bank criteria.
* At least 3 months incidence of typical freezing of gait (FOG) symptoms defined as the inability to move the feet despite the intention to walk including at least one of the following FOG patterns: start hesitancy, freezing at making turns or when passing through a doorway, spontaneous freezing during continued walking, or freezing of gait related to a simultaneous mental or physical activity.
* Freeze at least once per week (minimum score of 2 on item 3 of the FOG-Q) for at least 2 seconds (minimum score of 1 on item 4 of FOG-Q).
* Willing to attend assessment visits in the practically defined Off state having withdrawn from dopaminergic therapy: L-dopa preparations from midnight, Dopamine Agonists/Monoamine Oxidase-B Inhibitor for 36 hours prior to visit. Patients with device assisted therapies (i.e. Deep Brain Stimulation, L-dopa intestinal gel or subcutaneous apomorphine) to withdraw therapy for a minimum 30 minute period (maximum 2 hours) to achieve their clinically agreed Off state.
* Unless confirmed to be azoospermic (vasectomized or secondary to medical cause), males must agree to use a male condom from Day 1 throughout the study when having penile-vaginal intercourse with a woman of childbearing potential who is not currently pregnant. Men with a pregnant or breastfeeding partner must agree to remain abstinent from penile-vaginal intercourse or use a condom during each episode of penile-vaginal penetration until after the Follow-Up Visit.
* Females of childbearing potential (i.e., not postmenopausal or surgically sterile) who have a male partner must have a negative serum pregnancy test result and must agree to one of the following from start of Screening through 30 days after the last study medication administration: use a reliable method of birth control, or monogamous relationship with a male partner of confirmed sterility, or practice complete abstinence.
* Females of non-childbearing potential may be enrolled if it is documented that they are postmenopausal.
* Body weight greater or equal to 50 kg and body mass index (BMI) between 18 and 35 kg/m2, inclusive at Screening.
* Stable medical conditions for 3 months prior to Screening visit (e.g., controlled hypertension, dyslipidemia).
* Willing to follow the protocol requirements and comply with protocol restrictions.
* Capable of providing informed consent and complying with study procedures (completion of self-assessment rating scales and use of wearable devices). Subjects who are unable to provide consent may use a Legally Authorized Representative.

Exclusion Criteria:

* Poorly controlled hypertension despite lifestyle modifications and/or pharmacotherapy.
* Clinical signs indicating syndromes such as corticobasal degeneration, supranuclear gaze palsy, multiple system atrophy, chronic traumatic encephalopathy, signs of frontal dementia, history of stroke, head injury or encephalitis, cerebellar signs, early severe autonomic involvement, or Babinski sign.
* Current evidence or history in past two years of epilepsy, focal brain lesion, head injury with loss of consciousness or meeting DSM-IV diagnostic criteria for psychotic disorders, such as Schizophrenia or Bipolar Disorder, or have unstable concomitant psychiatric symptomatology.
* Evidence of any significant clinical disorder or laboratory finding (or in the case of potassium levels below normal range) that renders the participant unsuitable for receiving an investigational drug.
* History of malignant disease, including solid tumors and hematologic malignancies (except basal cell and squamous cell carcinomas of the skin that have been completely excised and are considered cured).
* Any clinically significant illness or disease as determined by medical and surgical history, physical examination, 12-lead electrocardiogram (ECG) and clinical laboratory assessments conducted at Screening.
* Clinically significant abnormalities of ECG, including QTcF > 450 ms, for males and QTcF > 470 ms for females, and/or heart rate < 50 beats per minute, or evidence of clinically significant bundle branch blocks, as indicated by 12-lead ECG.
* Calculated creatinine clearance of ≤70 mL/min according to the Cockcroft-Gault equation.
* Current use of any prohibited prescription medication, over-the-counter medication, or herbal supplements/products.
* Prior treatment with any investigational drug ≤90 days prior to dosing (Day 1), or ≤5 half-lives of the drug (whichever is longer), or current enrollment in any other study treatment or disease study except for observational studies.
* Known or suspected alcohol or substance abuse within the past 12 months.
* Suicidal ideation with actual intent or plan ("Yes" answer on the Columbia-Suicide Severity Rating Scale (C-SSRS) ideation items 4 or 5) within 3 months prior to study Screening.
* Current infection with severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2).
* Contraindications to wearing the BioStamp digital device sensors, which include but are not limited to implanted pacemakers, defibrillators, or other active implantable devices, and known allergies.
* Known hypersensitivities to adhesives or hydrogel.
* Females who are breastfeeding.
* Any other reason for which the PI considers it is not in the best interest of the participant to undertake the study.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-06 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Gait as Captured by Video Recordings | Days 1 and 14 of each Treatment Period (two 14-day periods)
  Subjects are requested to get up from a chair, walk to a square box shape taped to the floor five meters ahead and complete both a left and a right turn. Freezing of Gait (FOG) is tagged in the video at any point when a participant makes a sudden and involuntary cessation of normal progression of the feet through the task. The percentage time spent with FOG will be calculated by summing all FOG episodes and dividing by the total time to complete the task.

SECONDARY OUTCOMES:
Freezing of Gait Symptoms | Screening, Days 1 and 14 of each Treatment Period (two 14-day periods)
  The Freezing of Gait Questionnaire (FOG-Q) is an assessment of FOG severity. The FOG-Q consists of six items. Responses to each item use a 5-point interval scale ranging from 0, absence of symptoms to 4, most severe stage. The total score is calculated as the sum of the individual items and ranges from 0 to 24 with a higher score indicating more severe FOG.
Change from Baseline in CANTAB Reaction Time Task | Screening, Days 1 and14 of each Treatment Period (two 14-day periods)
  Measures changes in cognition by testing psychomotor speed (selecting a flashing circle on a touch tablet screen as quickly as possible).
Change from Baseline in CANTAB Paired Associates Learning Test | Screening, Days 1 and14 of each Treatment Period (two 14-day periods)
  Measures changes in cognition by testing attention (remembering the location of an abstract pattern on a touch tablet screen).
Change from Baseline in CANTAB Verbal Recognition Test | Screening, Days 1 and14 of each Treatment Period (two 14-day periods)
  Measures changes in cognition by testing memory (recall of 18 words flashed onto a touch tablet screen).
Digital wearable device (BioStamp) | Screening, Days 1-14 of each Treatment Period (two 14-day periods)
  A wireless device that measures physical activity and sleep (in hours/minutes) while at home

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Director — CuraSen Therapeutics, Inc.
Locations (1):
- The University of Sydney, Sydney, New South Wales, Australia